CLINICAL TRIAL: NCT01907958
Title: A Multicentre Study to Evaluate the Management of Microalbuminuria in Hypertensive Patients With Type 2 Diabetes: Improving Clinical Practice
Brief Title: Management of Albuminuria in Hypertensive Diabetics
Acronym: CLINPRADIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medpharmgene, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLINPRADIA
Record Dates: First submitted 2013-07-18; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Microalbuminuria; Hypertension; Type 2 Diabetes
Keywords: Microalbuminuria; Hypertensive; Diabetics; urine albumin
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — urine whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Multicenter stepped wedge cluster randomized trial of family practice clinics in Quebec and Ontario comparing the effect of introducing a Point of Care testing (POCT) for urine albumin to usual practice on quality of care in hypertensive patients with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years and older and able to visit the study sites every 3 months
* T2D patients with ongoing anti-diabetic therapy for at least 5 years
* Uncontrolled hypertension according to 2012 CHEP recommendations for management of hypertension in diabetic patients ( i.e. BP> 130/80 mmHg)
* Able and agreeing to provide informed consent.

Exclusion Criteria:

* Type 1 diabetes patients
* Ongoing therapy with perindopril,
* Known hypersensitivity or allergies to ACEI or sulfonamide derivatives,
* A history of angioedema related or not to previous treatment with ACEI,
* Impaired renal function defined as serum creatinine levels > 177 µmol/L, eGFR <30 mL/min,
* Hyperkalemia or hypokalemia,
* Severe hepatic impairment,
* Use of non-antiarrhythmic agents causing torsade de pointes,
* Pregnant or lactating women, or who are planning to become pregnant,
* Any conditions which may impact on participation according to treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years and older Uncontrolled blood pressure Type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Stabilisation or improvement of urine albumin excretion status by at least one stage | 1 year

SECONDARY OUTCOMES:
Microalbuminuria (or further stages of CKD) after 12 months | 12 months

OTHER OUTCOMES:
Demographics, medical history and medication Diabetes and hypertension status Blood pressure measurements | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medpharmgene, Montreal, Quebec, Canada